CLINICAL TRIAL: NCT04624282
Title: Metabonomics Study of Chronic Gastritis and Gastric Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Hanyuehua, Chief physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: I2020001797
Record Dates: First submitted 2020-10-19; First posted 2020-11-10 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with chronic superficial gastritis: Patients with chronic superficial gastritis
  Interventions: Diagnostic Test: different diseases
- Patients with chronic atrophic gastritis: Patients with chronic atrophic gastritis
  Interventions: Diagnostic Test: different diseases
- Patients with gastric carcinoma: Patients with gastric carcinoma
  Interventions: Diagnostic Test: different diseases

INTERVENTIONS:
Diagnostic Test: different diseases — Patients will be divided into three groups, including chronic superficial gastritis ,chronic atrophic gastritis and gastric carcinoma.

SUMMARY:
The pathogenetic mechanisms of chronic gastritis and gastric carcinoma are different. Whether metabonomics play a role in the development of chronic gastritis and gastric cancer is still a question. So the investigators want to clarify this question by this subject.

DETAILED DESCRIPTION:
This project was an untargeted metabolomics study using liquid chromatography coupled with mass spectrometry (LC-MS) in patients with chronic gastritis and gastric carcinoma. The experimental procedures mainly include sample collection, metabolite extraction, LC-MS/MS detection, data analysis, etc.The goal of this study is to identify and (relatively) quantify as many metabolites in biological systems as possible, so as to reveal the overall metabolite information to the maximum extent. Metabolomics aims to investigate the changes of metabolites in gastric tissues in patients with chronic gastritis and gastric carcinoma, and to study the biological processes in which these metabolites participate by screening the different metabolites in the different groups, and to reveal the mechanism of life activities in which they involved in.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic superficial gastritis and chronic atrophic gastritis
* Patients with gastric carcinoma

Exclusion Criteria:

* Patients with history of surgery
* Patients with severe heart disease,lung disease or kidney disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll patients with chronic superficial gastritis, chronic atrophic gastritis or gastric carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Metabonomic difference in patients with chronic gastritis and gastric carcinoma | six months
  1.The different levels of metabolites in gastric tissues in patients with chronic gastritis and gastric carcinoma. 2. The common change model of metabolites in gastric carcionoma compared with chronic gastritis.

SECONDARY OUTCOMES:
Association of different metabolic substances and disease results in chronic gastritis and gastric carcinoma | six months
  The researchers want to reveal the relationship between different metabolic sustances and disease result in patientswith chronic gastritis and gastric carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehua Han, Dr., Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang university, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No